CLINICAL TRIAL: NCT04874480
Title: Phase I Study of Tegavivint (BC-2059) in Patients With Relapsed and Refractory Leukemias
Brief Title: Tegavivint for the Treatment of Relapsed or Refractory Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0616; NCI-2021-03253 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0616 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-05-02; First posted 2021-05-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Leukemia; Refractory Leukemia
MeSH Terms: conditions — Leukemia | interventions — Decitabine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tegavivint, decitabine) (Experimental): PART I: Patients receive tegavivint IV over 4 hours on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  PART II: Patients receive tegavivint IV over 4 hours on days 1, 8, 15, and 22 and decitabine IV over 30-60 minutes on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Drug: Tegavivint

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Tegavivint — Given IV
  Other Names: BC 2059; BC-2059; BC2059; Tegatrabetan

SUMMARY:
This phase I trial is to find out the best dose and side effects of tegavivint in treating patients with leukemia that has come back (relapsed) or does not response to treatment (refractory). Tegavivint may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving tegavivint in combination with decitabine may help control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of tegavivint in patients with relapsed and refractory acute myeloid leukemia (AML). (Phase I dose escalation) II. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of tegavivint combined with decitabine in patients with relapsed and refractory acute myeloid leukemia (AML). (Combination cohort)

SECONDARY OBJECTIVES:

I. To assess the safety profile of tegavivint as characterized by adverse event (AE) type, severity, timing and relationship to study drug, as well as laboratory abnormalities in the first and subsequent treatment cycles. (Phase I dose escalation) II. To explore the efficacy (complete remission [CR], complete remission without blood count recovery [CRi], or partial remission [PR], of tegavivint as a single-agent in patients with relapsed/refractory (R/R) AML. (Phase I dose escalation) III. To assess overall survival (OS), and disease-free survival (DFS) in patients with R/R AML treated with tegavivint. (Phase I dose escalation) IV. To assess the duration of disease control defined as first date of disease control identified (either CR/CRi, PR or SD) until the date of progression. (Phase I dose escalation) V. To explore biomarkers of response and resistance in patients with R/R AML treated with tegavivint. (Phase I dose escalation) VI. To assess the safety profile of tegavivint in combination with decitabine as characterized by adverse event (AE) type, severity, timing and relationship to study drug, as well as laboratory abnormalities in the first and subsequent treatment cycles. (Combination cohort) VII. To explore the efficacy (complete response [CR], complete response without blood count recovery [CRi], or partial response [PR], of tegavivint in combination with decitabine in patients with R/R AML. (Combination cohort) VIII. To assess overall survival (OS), and disease free survival (DFS) in patients with R/R AML treated with tegavivint + decitabine. (Combination cohort) IX. To assess the duration of disease control defined as first date of disease control identified (either CR/ CRi, PR or SD) until the date of progression. (Combination cohort) X. To explore biomarkers of response and resistance in patients with R/R AML treated with tegavivint + decitabine. (Combination cohort)

OUTLINE: This is a dose-escalation study.

PART I: Patients receive tegavivint intravenously (IV) over 4 hours on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PART II: Patients receive tegavivint IV over 4 hours on days 1, 8, 15, and 22 and decitabine IV over 30-60 minutes on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of histologically confirmed relapsed or refractory (R/R) acute myeloid leukemia for which no available standard therapies are indicated or anticipated to result in a durable response
* Age >= 18 years
* Patients must not have had leukemia therapy for 14 days prior to starting tegavivint (BC-2059). However, patients with rapidly proliferative disease may receive hydroxyurea as needed until 24 hours prior to starting therapy on this protocol and during the first cycle of study
* Bilirubin =< 2.5 mg/dL
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN) - or =< 5 x ULN if related to leukemic involvement
* Creatinine =< 1.5 x ULN
* Known cardiac ejection fraction of > or = 45% within the past 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial
* Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol

Exclusion Criteria:

* Pregnant women are excluded from this study because the agent used in this study has the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided
* Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient with documented hypersensitivity to any of the components of the therapy program
* Patients with active, uncontrolled central nervous system (CNS) leukemia will not be eligible
* Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use at least 1 form of barrier birth control (such as condom) prior to study entry and for the duration of study participation
* Prior treatment with tegavivint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Adverse events will be tabulated with frequency and percentage by grade, attribution to treatment, and by dose level/schedule.
Response rate | Up to 2 years
  Response rate will be estimated alone with 95% confidence interval.
Overall survival | From date of treatment start until date of death due to any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method.
Disease free survival | From date of complete response (CR), or complete remission without blood count recovery (CRi) until the date of first objective documentation of disease-relapse or death, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method.
Duration of disease control | Up to 2 years
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org